CLINICAL TRIAL: NCT00074802
Title: CBT Augmentation of Paroxetine for Social Anxiety
Brief Title: Adding Cognitive Behavioral Therapy to Drug Treatment for Social Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH064481 (NIH); R01MH064481 (NIH); DSIR 83-ATAS; R01MH064726 (NIH); GSK ID: 101618 (Other: GlaxoSmithKline)
Record Dates: First submitted 2003-12-19; First posted 2003-12-22 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Social Anxiety Disorder
Keywords: Social Phobia
MeSH Terms: conditions — Phobia, Social | interventions — Paroxetine; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Open trial of paroxetine (Phase 1) followed by randomization to either continued paroxetine or continued paroxetine plus cognitive behavioral therapy (Phase 2) for patients showing partial response to paroxetine in Phase 1.
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators were unaware of randomized condition in the augmentation phase (Phase 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paroxetine Continuation (Experimental): Participants who showed only partial response to paroxetine in Phase 1 will receive continued treatment with paroxetine for 16 additional weeks.
  Interventions: Drug: Paroxetine
- Paroxetine with CBT Augmentation (Experimental): Participants who showed only partial response to paroxetine in Phase 1 will receive continued treatment with paroxetine plus cognitive behavioral therapy (CBT) for 16 additional weeks.
  Interventions: Drug: Paroxetine; Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Drug: Paroxetine — Treatment with paroxetine will consist of an immediate release, flexible dosage of 20 to 50 mg per day.
  Other Names: Paxil
Behavioral: Cognitive behavioral therapy (CBT) — CBT will consist of 16 weekly treatment sessions.
  Arms: Paroxetine with CBT Augmentation

SUMMARY:
This study will examine whether the addition of cognitive behavioral therapy can improve the efficacy of the medication paroxetine (Paxil®) in treating individuals with social anxiety disorder. Patients with social anxiety disorder will undergo a 12-week open trial with paroxetine. Those who complete the open trial having achieved only partial response will be randomized to receive cognitive behavioral therapy (CBT) in addition to paroxetine or to continue on paroxetine alone for an additional 16 weeks.

DETAILED DESCRIPTION:
Social anxiety disorder is a prevalent and disabling condition for which effective long-term treatments need to be identified. Paroxetine is effective in treating the acute symptoms of social anxiety, but many patients achieve less than optimal response. CBT has also been effective in treating social anxiety disorder; thus,it may also be effective in augmenting paroxetine response. This study will examine the effects of paroxetine treatment alone and in combination with CBT among patients who achieve less than optimal response after an open trial with paroxetine.

Participants in this study will receive paroxetine for 12 weeks (Phase 1). After 12 weeks, participants who have completed this open trial but have achieved some but less than optimal response will move forward to Phase 2. To be eligible to move forward to Phase 2, patients must have achieved at least a 10% improvement in their open-trial Liebowitz Social Anxiety Scale Scores (LSAS) but still have an LSAS score of 30 or greater. Patients meeting these criteria will be randomly assigned to either add weekly sessions of CBT to their treatment or to continue taking paroxetine alone for another 16 weeks. Social anxiety symptoms, rates of response and remission, fear of negative evaluation, disability and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders, Fourth edition (DSM-IV) criteria for generalized social phobia
* Willing and able to give written informed consent
* English-speaking

Exclusion Criteria:

* Prior or current diagnosis of schizophrenia, schizoaffective disorder, organic mental disorder, bipolar disorder, or antisocial, schizotypal, and schizoid personality disorders
* Suicidal thoughts
* History of failed paroxetine treatment of at least 6 weeks' duration at adequate doses or a history of failed outcome of a previous adequate trial of CBT
* Clinically significant and/or unstable medical disease
* Pregnancy or breast-feeding. Women of childbearing potential will be required to sign a statement indicating their intention to avoid pregnancy during the study through the use of an effective method of contraception.
* Alcohol or substance abuse or dependence within the past 3 months. Patients with a positive drug screen but no substance abuse disorder will be eligible for the study, provided they have not met criteria for abuse/dependence within the last 6 months and provide two clean urine samples 2 weeks apart.
* Current or past history of seizure disorder (except febrile seizure in childhood)
* Conditions that contraindicate the use of paroxetine
* Inability to tolerate or unwillingness to accept a drug-free period of 4 weeks for monoamine oxidase inhibitors (MAOIs) or fluoxetine and 2 weeks for other selective serotonin reuptake inhibitors (SSRIs), neuroleptics, antidepressants, benzodiazepines, mood stabilizers, buspirone, beta-adrenergic blockers, or other psychotropic drugs prior to beginning the study
* Currently receiving psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Heimberg, PhD, Principal Investigator — Adult Anxiety Clinic of Temple University; Michael Liebowitz, MD, Principal Investigator — New York State Psychiatric Institute Anxiety Disorders Clinic
Locations (2):
- United States (2):
  - New York State Psychiatric Institute Anxiety Disorders Clinic, New York, New York
  - Adult Anxiety Clinic of Temple University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in 2003 at the Adult Anxiety Clinic of Temple University and the Anxiety Disorders Clinic of the New York State Psychiatric Institute. 150 patients with Generalized Social Anxiety Disorder were enrolled in Phase I of the study (open treatment with the selective serotonin reuptake inhibitor paroxetine).
Pre-assignment Details: Among the 150 patients enrolled in Phase I, a total of 61 patients began Phase II These patients were classified as partial responders at week 12 (LSAS>29 but at least 10% improvement in LSAS score), and were therefore randomized to receive 16 weeks of continued treatment with paroxetine with or without CBT.
Period: Overall Study
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Started (Patients included here were the subset of enrollees completing the open trial as partial responders.) | 29 | 32
Completed | 20 | 25
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Population: Patients included here were the subset of enrollees completing the open trial as partial responders.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.38 (12.30) | 32.22 (9.73) | 33.72 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 19 | 24 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 8 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10
Liebowitz Social Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The Liebowitz Social Anxiety Scale is a 24-item clinician-administered measure, which provides 0-3 ratings for anxiety and avoidance of social and performance situations. Anxiety and avoidance ratings are summed across items, yielding a range of scores from 0-144, with higher scores representing greater severity of social anxiety symptoms.
  units on a scale | 49.45 (19.23) | 44.63 (13.60) | 46.92 (16.55)
Social Interaction Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — The Social Interaction Anxiety Scale is a 20-item self-report measure of anxiety experienced while interacting in dyads or groups. Items are rated on a 0-4 scale, yielding a range of scores from 0-80, with higher scores representing greater anxiety.
  units on a scale | 39.30 (11.08) | 35.43 (12.35) | 37.19 (11.85)
Social Phobia Scale [Mean (Standard Deviation); unit: units on a scale] — The Social Phobia Scale is a 20-item self-report measure of anxiety experienced when being observed by others. Items are rated on a 0-4 scale, yielding a range of scores from 0-80, with higher scores representing greater anxiety.
  units on a scale | 20.04 (11.87) | 17.43 (10.85) | 18.62 (11.29)
Brief Fear of Negative Evaluation Scale [Mean (Standard Deviation); unit: units on a scale] — The Brief Fear of Negative Evaluation Scale is a 12-item self-report measure of concern about negative evaluation by others. Items are rated on a 1-5 scale, yielding scores ranging from 12-60, with higher scores indicating greater fear of negative evaluation.
  units on a scale | 26.20 (7.34) | 21.83 (6.41) | 23.82 (7.13)
Liebowitz Self-Rated Disability Scale [Mean (Standard Deviation); unit: units on a scale] — The Liebowitz Self-Report Disability Scale is an 11-item self-report measure of the degree to which one's emotional problems limit one's ability to function in a variety of domains. Items are rated on a 0-3 scale of severity, and 10 of the 11 items (choosing either school or work as one area and omitting the other) are summed to produce a total score, ranging from 0-30. Higher scores represent greater disability.
  units on a scale | 8.42 (4.56) | 6.58 (4.40) | 7.42 (4.52)
Quality of Life Inventory [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life Inventory is a 16-item self-report measure of life satisfaction. Each item is rated for importance (0-2) and satisfaction (-3 to +3), and these ratings are multiplied, summed, and divided by the number of non-zero entries to yield an average item score, which can range from -6 to +6. Higher scores represent a higher quality of life.
  units on a scale | 0.67 (1.65) | 0.31 (1.67) | 0.48 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale (LSAS)
Description: The LSAS is a 24-item clinician-administered measure, which provides 0-3 ratings for anxiety and avoidance of social and performance situations. Anxiety and avoidance ratings are summed across items, yielding a range of scores from 0-144, with higher scores representing greater severity of social anxiety symptoms. We examined amount of change from week 12 to week 28 as the primary outcome. Change was calculated as Week 12 score minus Week 28 score, so a positive score equals greater positive change.
Time Frame: Change measured from Week 12 to Week 28
Population: Data analysis was conducted via mixed-effects linear regression which allows use of data from patients with missing observations by using maximum likelihood estimation. The same holds true for all continuous outcome measures. However, mean change (and SDs) reported here is based on completed observations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
units on a scale | 7.77 (22.49) | 7.84 (17.15)
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Test type: Superiority; p = .267, Mixed Models Analysis; Mean Difference (Net) = -5.43, 95% CI 2-sided [-15.05 to 4.19]

2. Secondary Outcome: Clinical Global Impression Improvement Scale (CGI-I)
Description: The CGI-I is a 7-point clinician-administered scale measuring improvement in symptoms over time. Lower numbers represent greater improvement. We examined responder status (i.e., percent of patients receiving an endpoint, Week 28, rating of 1 or 2) as well as remission status (i.e., percent of patients receiving an endpoint, Week 28, rating of 1) as secondary outcomes.
Time Frame: Responder and remitter status measured at Week 28
Population: Responders (CGI-I=1 or 2). Remitters (CGI-I=1). Analyses based on Week 28 observations if available. if not, Week 20 or Week 12 observations were substituted. Fisher's Exact Test used for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
Participants
  Responder Status: Responder | 17 | 28
  Responder Status: Non-Responder | 12 | 4
  Remitter Status: Responder | 3 | 11
  Remitter Status: Non-Responder | 26 | 21
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Fisher's Exact Test used for analyses of responder status; Test type: Superiority; p = .018, Fisher Exact — Fisher's Exact Test used for analyses
Statistical Analysis 2: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Fisher's Exact Test used for analyses of remitter status; Test type: Superiority; p = .034, Fisher Exact — Fisher's Exact Test used for analyses

3. Secondary Outcome: Social Interaction Anxiety Scale (SIAS)
Description: The SIAS is a 20-item self-report measure of anxiety experienced while interacting in dyads or groups. Items are rated on a 0-4 scale, yielding a range of scores from 0-80, with higher scores representing greater anxiety. We examined amount of change at from week 12 to week 28 as a secondary outcome. Change was calculated as Week 12 score minus Week 28 score, so a positive score equals greater positive change.
Time Frame: Change measured from Week 12 to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
units on a scale | 3.43 (9.58) | 5.67 (11.55)
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Test type: Superiority; p = .0005, Mixed Models Analysis; Mean Difference (Net) = -3.21, 95% CI 2-sided [-5.02 to -1.39]

4. Secondary Outcome: Social Phobia Scale (SPS)
Description: The SPS is a 20-item self-report measure of anxiety experienced when being observed by others. Items are rated on a 0-4 scale, yielding a range of scores from 0-80, with higher scores representing greater anxiety. We examined amount of change at from week 12 to week 28 as a secondary outcome. Change was calculated as Week 12 score minus Week 28 score, so a positive score equals greater positive change.
Time Frame: Change measured from Week 12 to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
units on a scale | 2.75 (10.29) | 5.83 (8.59)
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Test type: Superiority; p = .0775, Mixed Models Analysis; Mean Difference (Net) = -5.61, 95% CI 2-sided [-11.84 to 0.62]

5. Secondary Outcome: Brief Fear of Negative Evaluation Scale (BFNE)
Description: The BFNE is a 12-item self-report measure of concern about negative evaluation by others. Items are rated on a 1-5 scale, yielding scores ranging from 12-60, with higher scores indicating greater fear of negative evaluation. We examined amount of change at from week 12 to week 28 as a secondary outcome. Change was calculated as Week 12 score minus Week 28 score, so a positive score equals greater positive change.
Time Frame: Change measured from Week 12 to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
units on a scale | 1.13 (4.59) | 3.91 (5.69)
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Test type: Superiority; p = .0006, Mixed Models Analysis; Mean Difference (Net) = -5.53, 95% CI 2-sided [-8.70 to -2.35] — Paroxetine+CBT > Paroxetine alone in BFNE change

6. Secondary Outcome: Liebowitz Self-Report Disability Scale (LSRDS)
Description: The LSRDS is an 11-item self-report measure of the degree to which one's emotional problems limit one's ability to function in a variety of domains. Items are rated on a 0-3 scale of severity, and 10 of the 11 items (choosing either school or work as one area and omitting the other) are summed to produce a total score, ranging from 0-30. Higher scores represent greater disability. We examined amount of change at from week 12 to week 28 as a secondary outcome. Change was calculated as Week 12 score minus Week 28 score, so a positive score equals greater positive change.
Time Frame: Change measured from Week 12 to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
units on a scale | 1.25 (3.30) | -0.02 (2.72)
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Test type: Superiority; p = .871, Mixed Models Analysis; Mean Difference (Net) = 0.20, 95% CI 2-sided [-2.16 to 2.55]

7. Secondary Outcome: Quality of Life Inventory (QOLI)
Description: The QOLI is a 16-item self-report measure of life satisfaction. Each item is rated for importance (0-2) and satisfaction (-3 to +3), and these ratings are multiplied, summed, and divided by the number of non-zero entries to yield an average item score, which can range from -6 to +6. We examined amount of change at from week 12 to week 28 as a secondary outcome. Change was calculated as Week 12 score minus Week 28 score, so a positive score equals greater positive change.
Time Frame: Change measured from Week 12 to Week 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
Number analyzed (Participants) | 29 | 32
units on a scale | 0.25 (1.24) | -0.35 (1.72)
Statistical Analysis 1: Comparison: Paroxetine Continuation vs Paroxetine With CBT Augmentation; Test type: Superiority; p = .949, Mixed Models Analysis; Median Difference (Net) = 0.41, 95% CI 2-sided [-11.95 to 12.76]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed from the beginning of the open trial phase of the study and throughout the randomized phase in which patients received paroxetine with or without CBT. Data presented in the Serious Adverse Events (SAE) and AE tables refer to events occurring during the randomized phase (Weeks 12, 16, 20, 24, and 28).
Description: The pharmacotherapist used a checklist to inquire about the presence of 29 potential adverse effects at each visit and rated the severity of each on a scale from 0 to 3 (none, mild, moderate, or severe). Any event with a rating greater than 0 reported at any of the visits listed above is included here.
Arm/Group | Paroxetine Continuation | Paroxetine With CBT Augmentation
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/32
Other Adverse Events (participants affected / at risk) | 29/29 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine Continuation (N=29) | Paroxetine With CBT Augmentation (N=32)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) — 24 year old female reported heavy menstrual bleeding. It was determined that the bleeding was likely related to polycystic ovarian syndrome. Bleeding returned to normal levels after initiation of hormone treatment. SAE unrelated to study meds.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine Continuation (N=29) | Paroxetine With CBT Augmentation (N=32)
Headache (General disorders) | 11 (25) | 11 (23)
Palpitations (General disorders) | 10 (29) | 5 (9)
Myalgia (General disorders) | 10 (20) | 2 (6)
Nausea (General disorders) | 11 (16) | 6 (10)
Vomiting (General disorders) | 4 (5) | 4 (5)
Sweating (General disorders) | 12 (37) | 4 (11)
Photophobia (General disorders) | 4 (15) | 3 (11)
Tachycardia (General disorders) | 8 (24) | 4 (6)
Bradycardia (General disorders) | 2 (8) | 2 (2)
Constipation (General disorders) | 15 (38) | 5 (9)
Diarrhea (General disorders) | 4 (14) | 4 (6)
Lightheadedness (General disorders) | 15 (30) | 9 (13)
Dry Mouth (General disorders) | 13 (24) | 8 (16)
Blurry Vision (General disorders) | 4 (13) | 2 (5)
Parathesias (General disorders) | 3 (5) | 3 (4)
Decreased Libido (General disorders) | 16 (51) | 18 (58)
Anorgasmia (General disorders) | 20 (73) | 18 (65)
Impaired Coordination (General disorders) | 3 (5) | 3 (7)
Fatigue (General disorders) | 14 (48) | 15 (41)
Nervousness (General disorders) | 14 (32) | 11 (30)
Insomnia (General disorders) | 10 (24) | 9 (17)
Tremor (General disorders) | 5 (11) | 7 (18)
Weight Gain (General disorders) | 19 (48) | 18 (52)
Weight Loss (General disorders) | 5 (8) | 7 (13)
Dermatitis (General disorders) | 6 (6) | 4 (7)
Urinary Congestion (General disorders) | 6 (19) | 6 (11)
Nasal Congestion (General disorders) | 7 (20) | 9 (12)
Rigidity (General disorders) | 7 (19) | 4 (4)
Somnolence (General disorders) | 16 (46) | 17 (49)

LIMITATIONS AND CAVEATS:
Limitations include the small size of the randomized sample and the lack of a placebo arm in the randomization phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No